CLINICAL TRIAL: NCT04818073
Title: Determinants of the Effectiveness of Robot-assisted Hand Movement Training
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of Idaho (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, David Reinkensmeyer, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 476; 2R01HD062744-06 (NIH)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Stroke, Ischemic; Cerebrovascular Accident (CVA)
Keywords: Rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomized single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Participants with undergo new FINGER robotic training with no physical assistance 3 times a week for a period of 3 weeks.
  Interventions: Device: New FINGER
- Group B (Experimental): Participants will undergo new FINGER robotic training with physical assistance 3 times a week for a period of 3 weeks.
  Interventions: Device: New FINGER
- Group C (Experimental): Participants will undergo new FINGER robotic training with physical assistance and proprioceptive exercises 3 times a week for a period of 3 weeks.
  Interventions: Device: New FINGER

INTERVENTIONS:
Device: New FINGER — New FINGER exoskeleton is a robotic device that can provide assistance and resistance to thumb and finger movement

SUMMARY:
The investigators would like to investigate the effectiveness of somatosensory training for robot-assisted hand motor rehabilitation after stroke.

DETAILED DESCRIPTION:
From previous studies, the investigators learned that stroke survivors with impaired finger proprioception did not achieve as large a functional benefit from robotic finger training. For this study, the investigators would like to determine if and the extent of finger proprioception can be improved through targeted robotic proprioceptive training combined with robotic finger movement training. The investigators would also include imagining studies via Electroencephalogram (EEG) and other baseline predictors to provide insight to determine who responds best to proprioceptive training.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years
* Suffered from a single ischemic stroke (radiologically confirmed) at least 6-months prior to enrollment
* An ability to score at least 3 blocks on the Box and Block Test

Exclusion Criteria:

* A substantial decrease in alertness, language reception or attention
* Pregnant or lactating
* Advanced liver, kidney, cardiac or pulmonary disease
* Plan to alter any current participation in other rehabilitation therapy in the time period of the study
* A terminal medical diagnosis consistent with survival < 1 year
* Coexistent major neurological disease
* Coexistent major psychiatric disease
* A history of significant alcohol or drug abuse in the prior 3 years
* Current enrollment in another study related to stroke or stroke recovery
* Any other medical contraindication to participation in this study evaluated by our team physician.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Box and Blocks Test | From baseline to 1-month post intervention
  We compare the change of Box and Block Test scores from baseline evaluation to 1-month post intervention. Participants are instructed to move as many blocks as possible, one at a time, from one compartment in a box to a second compartment over a divider for a period of 60 seconds; each block that is moved is counted, and multiple blocks moved at the same time are counted as a single block. The higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Fugl-Meyer Motor Assessment of the Upper Extremity | From baseline to 1-month post intervention
  We will measure the change of the Fugl-Meyer Motor Assessment scores from the baseline evaluation to 1-month post intervention. Fugl-Meyer is a 66-point scale measuring the movement pattern of upper extremities. The higher scores indicate a better outcome.
Motor Activity Log | From baseline to 1-month post intervention
  We will measure the change of the Motor Activity Log (MAL) mean scores from the baseline evaluation to 1-month post intervention. The Motor Activity Log is a 30 questionnaire that collect subjective measure of an individual's real life functional upper limb performance. The higher scores indicate a better outcome.
Changes in finger proprioception measured using the Crisscross Assessment. | From baseline to 1-month post intervention
  We will measure the change in finger proprioception scores from the baseline evaluation to 1-month post intervention. Finger proprioception is measured by using the FINGER Crisscross Assessment which we slowly move the index and middle fingers with the FINGER robot past each other without any visual input. We then ask study participants to press a key when they feel the fingers are overlapped. Finger proprioception is measured by the error which will be quantified as the mean magnitude of finger separation error at the metacarpal joint when the key is pressed. The lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David Reinkensmeyer, Ph.D, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowe JB, Chan V, Ingemanson ML, Cramer SC, Wolbrecht ET, Reinkensmeyer DJ. Robotic Assistance for Training Finger Movement Using a Hebbian Model: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2017 Aug;31(8):769-780. doi: 10.1177/1545968317721975. PMID 28803535
- [Background] Ingemanson ML, Rowe JB, Chan V, Wolbrecht ET, Cramer SC, Reinkensmeyer DJ. Use of a robotic device to measure age-related decline in finger proprioception. Exp Brain Res. 2016 Jan;234(1):83-93. doi: 10.1007/s00221-015-4440-4. Epub 2015 Sep 16. PMID 26378004